CLINICAL TRIAL: NCT04484792
Title: Green Tea Mouthwash on Generalized Plaque- Induced Gingivitis: A Randomized Controlled Clinical Trial
Brief Title: Green Tea Mouthwash on Generalized Plaque- Induced Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Alhanouf M. AlRehaili, Principal Investigator, Taibah University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: TUCDREC/20181112/AlRehaili
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Plaque Induced Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Other: green tea mouthwash
- Group B (Experimental)
  Interventions: Other: green tea mouthwash
- Group C (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: green tea mouthwash — green tea bags in 100 ml warm water for 5 min
  Arms: Group A
Other: green tea mouthwash — , in Group B its prepared by soaking tea bags in 100 ml hot water followed by ice addition.
  Arms: Group B
Other: placebo — Plain water
  Arms: Group C

SUMMARY:
This investigation will study the effect of green tea mouthwash as an adjunctive therapy to mechanical treatment on gingival health, and whether it has any side effects. This study also aims at increasing the awareness among health professionals and the community regarding the benefits of natural herbal products such as green tea on oral health, opposed to common chemical products. This may provide an efficient alternative for people who are sensitive to certain chemical products or who have limited sources of income and cannot afford expensive treatment of dental problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the clinics at the Taibah University Dental College and Hospital (TUDCH)
* Age from 18 - 35 years
* Generalized plaque-induced gingivitis (GBI > 85%)

Exclusion Criteria:

* Patients with any systemic diseases
* Patients under regular medication (e.g. Contraceptives, Hormone- Replacement Therapy)
* Pregnant or breast-feeding patients
* Smokers
* Periodontitis patients
* Patients who received any form of periodontal therapy within the last 6 months
* Patients who were under antibiotic therapy the past month
* Patients using regular mouthwash or other chemical plaque control agents (e.g. Miswak) except for regular toothpaste (Note: toothpastes with specific anti-inflammatory properties are excluded)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
plaque control record | over 27 days
gingival bleeding index | over 27 days

CONTACTS AND LOCATIONS:
Locations (1):
- Taibah University, Al Madīnah, Saudi Arabia